CLINICAL TRIAL: NCT00011622
Title: Maternal Glucose Measurement in Pregnancy Using a Continuous Ambulatory Subcutaneous Monitor
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Other Study IDs: NCRR-M01RR02558-0158
Record Dates: First submitted 2001-02-22; First posted 2001-02-26 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Device: Continuous ambulatory subcutaneous glucose monitor

SUMMARY:
This proposal is a pilot study to describe the variations of blood sugar in pregnant women with various degrees of glucose intolerance, and how they relate to standardized meals. Blood sugar control during pregnancy is important to prevent complications for the newborn. The variation and timing of the blood sugar measurements in gestational diabetics and how this relates to the baby's outcome is controversial. We will use an FDA approved device called Minimed Glucose Continuous Monitor, which is used in clinical practice for certain diabetics. It is very small, similar to a beeper, and is connected to the patient through a small plastic catheter subcutaneously. This measures blood sugar every five minutes for a total of 288 readings a day with minimum discomfort. The hypothesis of this study is that use of the Minimed glucose monitor will provide information about variations of blood sugar in gestational diabetics that is missed by capillary glucose monitors.

Our conclusions will allow us to compare blood glucose trends among the groups. After the data is analyzed in this pilot study, we plan to design a bigger study involving more subjects to study the impact of the blood sugar variations in the outcome of the newborn, and to obtain generalizable results for the population in general.

DETAILED DESCRIPTION:
We will coordinate the study through the CRC. The women will have to come in only twice, to have the monitor placed and then taken off three days later. A blood sample will be collected at each visit. Meals and snacks will be provided for each day of the study, specially packaged, to supply an equivalent amount of calories for each subject. These will meet the nutritional requirements for both the mother and the fetus. Women will do separate fingerstick blood sugar measurements using a capillary glucometer four times a day, to ensure the accuracy of the sensor's readings.

ELIGIBILITY:
1. Inclusion Criteria

* Pregnant women, between 28 and 36 weeks of gestation. Gestational age will be determined by a combination of the date of the last menstrual period and ultrasound, done during the first or second trimester of pregnancy.
* Previous glucose challenge test and if abnormal, an oral glucose tolerance test.
* Body mass index (BMI) between 25 and 30 Kg/m2.
* Gestational diabetes in a previous pregnancy, if glucose between pregnancies was normal.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Medical School, Houston, Texas, United States